CLINICAL TRIAL: NCT05577923
Title: Exploring Whether Disease-free Intervals Can Guide Endocrine Combined Targeted Therapy for ER+/HER2+ Advanced Breast Cancer (T-sunflower)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUSCC-T-sunflower
Record Dates: First submitted 2022-08-18; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; pyrotinib; dalpiciclib; Fulvestrant

STUDY DESIGN:
Intervention Model Description: Depending on the DFI, the subjects will be divided into four groups, namely T0, TS(≤2 years), TM(2-5 years), and TL(≥5 years). All subjects will receive the same treatment regimen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T-sunflower group (Experimental): Patients will be treated with Trastuzumab, Pyrotinib, Dalpiciclib plus Fulvestrant.
  Interventions: Drug: Trastuzumab; Drug: pyrotinib; Drug: Dalpiciclib; Drug: fulvestrant

INTERVENTIONS:
Drug: Trastuzumab — 8 mg/kg loading dose IV, then 6 mg/kg IV, every 3 weeks
Drug: pyrotinib — Pyrotinib 320mg, PO daily, continuously
Drug: Dalpiciclib — Dalpiciclib will be given at the dose of 125 mg po q.d. x 21 every 4 weeks
Drug: fulvestrant — Fulvestrant will be given intramuscle at the dose of 500 mg every 4 weeks (with an additional 500 mg dose given two weeks after the initial dose.

SUMMARY:
This study is a prospective, single-arm, phase II clinical study for patients with ER+/HER2+ advanced breast cancer.

DETAILED DESCRIPTION:
Patients with ER+/HER2+ advanced breast cancer are planned to be enrolled. Patients will receive first-line endocrine therapy combined with anti-HER2 therapy. The main purpose is to evaluate whether disease-free intervals can guide first-line endocrine combined targeted therapy for ER+/HER2+ advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

Females ≥18 years and ≤ 75 years old;

* Histologically confirmed ER + / HER2- invasive breast cancer (specific definition: immunohistochemical detection of ER> 10% tumor cell positive is defined as ER positive, HER2 3+ or HER2 amplification followed by FISH detection);
* Stage IV breast cancer or recurrent metastatic breast cancer;
* Patients had received no previous chemotherapy or targeted therapy for metastatic disease
* At least one lesion (measurable and/or non-measurable) that has not previously received radiation therapy
* Normal heart function, normal ECG and LVEF ≥ 55%;
* Has adequate bone marrow function: absolute neutrophil count > 1.5x10ˆ9 /L; platelet count > 75x10ˆ9 /L, hemoglobin > 9g/dL;
* Has adequate liver function and kidney function: TBIL ≤1.5 times of the normal upper limit；ALT and AST ≤3 times of the normal upper limit；if liver metastases，then ALT and AST≤ 5 times of the normal upper limit；serum creatinine ≤1.5 times of the normal upper limit; Child-Pugh A/B（≤9 score）
* Participants voluntarily joined the study, has signed informed consent before any trial related activities are conducted, has good compliance and has agreed to follow-up.

Exclusion Criteria:

* Treatment with chemotherapy, radiotherapy, immunotherapy or surgery (outpatient clinic surgery excluded) for metastatic disease
* CNS metastases
* Significant cardiovascular disease(including congestive heart failure, angina pectoris, myocardial infarction or ventricular arrhythmia in the last 6 months);
* is pregnant or breast feeding;
* Malignant tumors in the past five years (except cured skin basal cell carcinoma and cervical carcinoma in situ).
* Positive test for human immunodeficiency virus
* Active hepatitis B or hepatitis C
* Rapid progression of the disease, researchers judge that endocrine combination targeted therapy is not suitable, including the number of liver metastases exceeding 10 or the maximum diameter of a single liver metastases ≥ 10 cm, symptomatic thoraco-ascites, etc.;
* Subjects with uncontrolled lung disease, severe infection, active gastrointestinal ulcer, coagulopathy, severe uncontrolled diabetes, connective tissue disease or inhibition of bone marrow function who cannot tolerate therapy;
* Current use or anticipated need for food or drugs that are known strong CYP3A4 (cytochrome P450 3A4) inhibitors or inducers.

  1. Strong CYP3A inhibitors, including, boceprevir, clarithromycin, conivaptan, delavirdine, indinavir, itraconazole, ketoconazole, lopinavir, mibefradil, miconazole, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, suboxone, telaprevir, telithromycin, voriconazole, and grapefruit, grapefruit juice or any product containing grapefruit.
  2. Strong CYP3A inducers, including carbamazepine, phenytoin, primidone, rifampin, rifapentin, and St. John's wort.
* Moderate infection occurs within 4 weeks before the first administration (e.g. intravenous drip of antibiotics, antifungal or antiviral drugs according to clinical criteria), fever of unknown origin occurs during the screening period/before the first administration.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
PFS | Randomization until the first occurrence of disease progression or death from any cause, which ever occurs first, through the completion of study (approximately 5 years)
  time to progressive disease (according to RECIST1.1)

SECONDARY OUTCOMES:
ORR | Randomization until the first occurrence of disease progression or death from any cause, which ever occurs first, through the completion of study (approximately 5 years)
  The proportion of participants whose best outcome is complete remission or partial remission (according to RECIST1.1)
CBR | Randomization until the first occurrence of disease progression or death from any cause, which ever occurs first, through the completion of study (approximately 5 years)
  the percentage of subjects with CR+PR+SD and last more than 24 weeks in all of the
DOR | Randomization until the first occurrence of disease progression or death from any cause, which ever occurs first, through the completion of study (approximately 5 years)
  Duration of whose best outcome is complete remission or partial remission (according to RECIST1.1)

CONTACTS AND LOCATIONS:
Overall Officials: zhimin U Shao, professor, Principal Investigator — Fudan University Shanghai Cancer Center Shanghai, China, 200032
Locations (1):
- Fudan University Shanghai Cancer Center Shanghai, China, 200032, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No